CLINICAL TRIAL: NCT04155164
Title: Effect of Metformin on Visual Function in Patients With Primary Open Angle Glaucoma: A Randomized Control Study
Brief Title: Effect of Metformin on Visual Function in Patients With Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019KYPJ130
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma; Metformin; Visual function
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and researchers are double-blind. After signing informed consent, subjects who meet the inclusion criteria will be randomly divided into the oral Metformin experimental group or the oral placebo control group at a ratio of 1:1. Random lists will be generated by independent statisticians. Randomized group will be sealed in a separate opaque envelope, showing only the research identification number. Participants and researchers (medical evaluators, outcome evaluators and data analysts) will be unaware of the grouping.
  During the period of treatment, if patient suffers from lactic acidosis, excessive ventilation, myalgia, the masking should be unveiled and his/her systematic and eye conditions should be assessed to choose the best treatment. The choice of remedial treatment plan is based on the consensus of doctors and patients. The changes of treatment methods and curative effect should be recorded in detail for future analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Participants will receive Metformin for 12 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Participants will receive placebo for 12 months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Metformin — Participants will receive Metformin at 1000mg for 12 months.
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebos — Placebo group will take Placebo at 1000mg for 12 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Metformin could prevent the progression of glaucoma in a safe and effective manner.

DETAILED DESCRIPTION:
Primary open-angle glaucoma (POAG) is a serious blinding disease characterized by irreversible damage to retinal ganglion cells (RGCs). At present, there is no effective treatment for the rescue of visual function loss caused by POAG.

Metformin is the classic first-line therapy for diabetes. Recently, it has been found that Metformin may have other beneficial effects such as promoting weight loss and reversing age-related neurodegeneration. Importantly, retrospective case-control studies found that there were associations between Metformin treatment and a reduction in the incidence of glaucoma. Specifically, diabetic patients treated by Metformin had a 25% lower risk to develop open-angle glaucoma. In addition, previous animal experiments have preliminarily shown that Metformin can play a neuroprotective role by activating AMPK kinase, regulating methylation levels and promoting ganglion cell survival. Therefore, the investigators hypothesize that Metformin can prevent visual function deterioration via rescuing retinal ganglion cells.

The main objective of this study is to assess the progression of visual field loss in patients with POAG after treatment with Metformin versus placebo. The secondary objectives include the followings: RNFL thickness, vision, cup/disk ratio, safety, and biochemical tests to determine the alteration of AMPK and methylation parameters associated to the use of Metformin.

Approximately 40 study subjects will be randomized in a 1:1 ratio to each treatment group. The treatment group will be assigned to the study intervention (oral Metformin) for 12 months while the placebo group will receive placebo containing fructose and starch for 12 months. Throughout the 12-month study period, progression of visual function and systematic safety examinations will be measured. At 18 months, there will be one additional follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years old;
* The baseline value of intraocular pressure ≤ 21 mmHg in either eye whether untreated or treated by ≤ 2 eye drops (laser or filtering surgery should be performed over 3 months).
* Over two times of experience of visual field examination (24-2 or 30-2 visual field examinations) in the past two years, or false positive/false negative ratio less than 33%;
* Diagnosed POAG by Glaucoma specialists from Zhongshan Ophthalmic Center with open angle, and impairment in optic disc or visual field in one or both eyes.
* Patient is at risk of glaucomatous progression, as determined by the documented presence of optic disc hemorrhage within 12 months in either eye, OR ≥2 of the following risk factors:
* Vertical cup-to-disc ratio >0.8 in one or both eyes
* Mean deviation in visual field worse than <10 dB in either eye (verified by the reading center)
* Pseudoexfoliation in either eye
* Family history (parent or sibling) of glaucoma
* Hypertension
* Systemic hypertension requiring medical treatment Migraine (defined by the International Headache Society with or without aura, Raynaud's syndrome, or both:
* The main organs are functioning normally and meet the following criteria:

  1. Blood sample should meet the following criteria: (no blood transfusion within 14 days) A. Hemoglobin (> 90g/L); B. Platelet count (>105*10e9/L)
  2. Biochemical and urinary examinations should meet the following criteria:

  <!-- -->

  1. . Urine bilirubin < 1.25 times ULN (Upper Limit of Normal);
  2. . ALT and AST < 2.5 times ULN;
  3. . CREA ≤ ULN;

Exclusion criteria:

* Secondary open-angle glaucoma (such as pigmentation syndrome, trauma, etc.) or angle-closure glaucoma.
* The best corrected visual acuity of either eye is less than 6/36;
* The mean derivation of visual field in either eye is less than - 22dB.
* Use of >2 topical (or any oral) IOP-lowering products at the baseline visit.
* Any ocular pathology in either eye that may have interfered with the ability to obtain visual field, disc imaging, or accurate IOP readings such as uveitis, refractive opacification;
* Eye drops such as neuroprotective therapies have been used in the past three weeks might affect this clinical study, for inclusion need 8 weeks of wash period.
* Pregnant or nursing women;
* Diabetes mellitus, definite impairment of liver and kidney function, or severe heart, liver or kidney diseases;
* In the last three months, ophthalmic surgery (including cataract surgery) has been performed
* Enrolled in other clinical study at the same time.
* Could not complete the study according to the requirements in this research .
* History of epilepsy or severe mental illness, including schizophrenia, bipolar disorder or severe depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Visual field | 0 months, 12 months
  to measure the change in visual field loss

SECONDARY OUTCOMES:
Changes in best corrected visual acuity (BCVA) | 0 months, 6 months, 12 months
  to measure the change in visual acuity
Changes in retinal RNFL thickness | 0 months, 6 months, 12 months
  to meausre the thickness of retinal RNFL by OCT
Changes in retinal cup/disk ratio | 0 months, 6 months, 12 months
  to measure the alterations in retina cup/disk ratio
Systemic safety as measured by presence of side effects listed on Metformin drug label as "severe" | 0 months, 6 months, 12 months
  These include:
  Infrequent side effects of Metformin (severe):Dyspnea;
  Rare side effects of Metformin (severe):Lactic acidosis; Hypoglycemia; Megaloblastic Anemia; Allergic reactions.
  The participants will be assessed for these side-effects at each follow-up ocular exam to confirm ocular and systematic safety of Metformin. Blood samples will be collected at 0 month, 6 months, and 12 months to value AMPK, methylation level and inflammatory responses. The Data Monitoring Committee for this study will also assess the safety of Metformin at different time points throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xialin Liu, Prof., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Xing Liu, Prof., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No